CLINICAL TRIAL: NCT02663531
Title: Retinal Neuro-vascular Coupling in Patients With Neurodegenerative Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OPHT-180515
Record Dates: First submitted 2015-12-21; First posted 2016-01-26 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease; Healthy
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mild cognitive impairment (Experimental): Patients with mild cognitive impairment
  Interventions: Device: DVA; Device: FDOCT; Device: Pattern ERG; Device: Optical Coherence Tomography
- Alzheimer Disease (Experimental): Patients with Alzheimer Disease
  Interventions: Device: DVA; Device: FDOCT; Device: Pattern ERG; Device: Optical Coherence Tomography
- Healthy (Experimental): Healthy volunteers
  Interventions: Device: DVA; Device: FDOCT; Device: Pattern ERG; Device: Optical Coherence Tomography

INTERVENTIONS:
Device: DVA
  Other Names: Dynamic Vessel Analyzer
Device: FDOCT
  Other Names: Fourier Domain Color Doppler Optical Coherence Tomography
Device: Pattern ERG
Device: Optical Coherence Tomography

SUMMARY:
Alzheimer´s disease (AD) in one of the most important causes of dementia and poses a considerable challenge in health care. Today, criteria for the diagnosis and the follow up of patients with AD mainly rely either on subjective tests or invasive methods. This limits the general applicability of the latter test for population screening and underlines the need for the identification of easily accessible tools for the identification of high-risk subjects. Because of its unique optical properties, the eye offers the possibility of the non-invasive assessment of both structural and functional alterations in neuronal tissue. As the neuro-retina is part of the brain, it does not come as a surprise that neuro-degenerative changes in the brain are accompanied by structural and possibly also functional changes in the neuro-retina and the ocular vasculature. The current study seeks to test the hypothesis that beside the known anatomical changes, also functional changes can be detected in the retina of patients with AD. For this purpose, flicker light induced hyperemia will be measured in the retina as a functional test to assess the coupling between neural activity and blood flow. Further, structural parameters such as retinal nerve fiber layer thickness and function parameters such as ocular blood flow and retinal oxygenation will be assessed and compared to age and sex matched controls.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for healthy subjects

* Men and women aged over 50 years
* Non-smokers
* Normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia < 6 Dpt

Inclusion criteria for patients with AD:

* Men and women aged over 50 years
* Normal ophthalmic findings, ametropia < 6 Dpt.
* Confirmed diagnosis of probable AD of mild to moderate degree defined as:

  1. Diagnosis of probable Alzheimer's disease based on the NINCDS/ADRDA criteria
  2. Assessing the severity of Alzheimer's disease of mild to moderate degree by the Mini Mental State Examination (MMSE). AD of mild to moderate degree has been confirmed if the MMSE score is in the range of 20 to 26 inclusive
* Hachinski Ischemia Scale is used to try and distinguish AD from multi-infarct dementia. A score of ≤ 4 suggests AD Informed consent capability
* Adequate visual and auditory acuity to allow neuropsychological testing and participation in the ocular blood flow measurements
* A potential participant has to be on stable doses of all medications he/she is taking because of consisting illnesses according to medical history (except AD therapy itself which will be recorded separately) for at least 30 days prior inclusion, if considered relevant by the investigator.

Inclusion criteria for patients with mild cognitive impairment:

* Men and women aged over 50 years
* Normal ophthalmic findings, ametropia < 6 Dpt.
* Diagnosis of probable mild cognitive impairment (MCI) defined as:

  1. memory complaint, corroborated by an informant
  2. abnormal memory function, documented by delayed recall of one paragraph from the Logical Memory II subtest of the Wechsler Memory Scale-Revised (cutoff scores: ≤8 for ≥16 years of education; ≤4 for 8 to 15 years of education; and ≤2 for 0 to 7 years of education [the maximum number of paragraph items possible to correctly recall is 25])
  3. normal general cognitive function, as determined by a clinician's judgment based on a structured interview with the patient and an informant (Clinical Dementia Rating [CDR]) and a Mini-Mental State Examination (MMSE) score greater than 26
  4. no or minimal impairment in activities of daily living (ADLs), as determined by a clinical interview with the patient and informant
  5. not sufficiently impaired, cognitively and functionally, to meet the NINCDS/ADRDA criteria, as judged by an experienced AD research clinician
* Hachinski Ischemia Scale is used to try and distinguish MCI from multi-infarct dementia. A score of ≤ 4 suggests MCI Informed consent capability
* Adequate visual and auditory acuity to allow neuropsychological testing and participation in the ocular blood flow measurements
* A potential participant has to be on stable doses of all medications he/she is taking because of consisting illnesses according to medical for at least 30 days prior inclusion, if considered relevant by the investigator.

Exclusion Criteria for patients:

* Presence or history of a severe medical condition other than cognitive impairment as judged by the clinical investigator
* Untreated Arterial hypertension
* History or family history of epilepsy
* Presence of any abnormalities preventing reliable measurements in the study eye as judged by the investigator
* Best corrected visual acuity < 0.5 Snellen
* Ametropia greater than 6 Dpt
* pregnancy or planned pregnancy
* Major psychiatric disorder (e.g. schizophrenia), if considered relevant by the investigator
* Significant neurological disease other than AD or MCI, if considered relevant by the investigator
* Alcoholism or substance abuse

Exclusion criteria for healthy volunteers:

* Presence or history of a severe medical condition as judged by the clinical investigator
* Untreated Arterial hypertension
* History or family history of epilepsy
* Presence of any abnormalities preventing reliable measurements in the study eye as judged by the investigator
* Family history of AD
* Best corrected visual acuity < 0.5 Snellen
* Ametropia 6 Dpt
* Pregnancy or planned pregnancy

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-09-27 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Flicker induced increase in retinal blood flow | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhöfer, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria